CLINICAL TRIAL: NCT06853535
Title: Precision Antiplatelet Therapy Guided by Platelet Aggregation Function in Patients With Acute Ischemic STROKE
Acronym: PATH STROKE C
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Fudan University (Other); Chengdu Medical College (Other)
Responsible Party: Principal Investigator, Jie Yang, Deputy Director of the Department of Neurology, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IITLX2025007
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Acute Ischemic Stroke; Clopidogrel Resistance
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ticagrelor (Experimental): Ticagrelor 90 mg should be administered as early as possible (within 12-24 hours after the loading dose).
  From Day 1 to Day 21 after enrollment: Patients shall receive dual antiplatelet therapy with oral ticagrelor 90 mg bid and aspirin 100 mg qd.
  From Day 22 to Day 90 after enrollment: Patients shall receive monotherapy with oral ticagrelor 90 mg bid.
  Interventions: Drug: The ticagrelor
- The Clopidogrel (Other): From the 1st to the 21st day, the patient should receive dual anti - platelet therapy with clopidogrel 75mg once a day (qd) combined with aspirin 100mg once a day (qd). From the 22nd to the 90th day, the patient should be given clopidogrel 75mg qd for anti - platelet treatment.
  Interventions: Drug: The Clopidogrel

INTERVENTIONS:
Drug: The ticagrelor — Ticagrelor 90 mg should be administered as early as possible (within 12-24 hours after the loading dose).
  From Day 1 to Day 21 after enrollment: Patients shall receive dual antiplatelet therapy with oral ticagrelor 90 mg bid and aspirin 100 mg qd.
  From Day 22 to Day 90 after enrollment: Patients shall receive monotherapy with oral ticagrelor 90 mg bid.
  Arms: The ticagrelor
Drug: The Clopidogrel — From the 1st to the 21st day, the patient should receive dual anti - platelet therapy with clopidogrel 75mg once a day (qd) combined with aspirin 100mg once a day (qd). From the 22nd to the 90th day, the patient should be given clopidogrel 75mg qd for anti - platelet treatment.
  Arms: The Clopidogrel

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of platelet aggregation function - guided precision anti - platelet therapy in patients with acute cerebral infarction. The main question it aims to answer is: among the cerebral infarction patients with possible clopidogrel resistance detected by platelet aggregation function tests, what is the efficacy and safety of using ticagrelor to replace the clopidogrel treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patients diagnosed with acute non-disabling ischaemic stroke or transient ischaemic attack (TIA) with moderate to high stroke risk in accordance with the WHO diagnostic criteria, defined as follows:

   * Acute non-disabling ischaemic stroke: NIHSS score ≤ 5 at enrollment;
   * TIA with moderate to high stroke risk: ABCD₂ score ≥ 4.
3. Time from symptom onset ≤ 48 hours. (Definition of symptom onset time: the interval from the last time the patient was observed in a normal state to the time of co-administration of clopidogrel 300 mg and aspirin 100 mg.)
4. MARADP ≥ 35% measured at 5-20 hours after the patient received antiplatelet therapy with co-administration of clopidogrel 300 mg and aspirin 100 mg within 48 hours of symptom onset.
5. Written informed consent signed by the patient or their legal representative.

Exclusion Criteria:

1. Imaging examinations suggestive of hemorrhagic stroke, hemorrhagic transformation, or other pathological cerebral disorders, such as vascular malformation, tumor, abscess, or other common non-ischemic cerebral diseases (e.g., multiple sclerosis).
2. Minor stroke/TIA induced by angioplasty or vascular surgery.
3. Routine electrocardiogram (ECG) suggestive of atrial fibrillation (AF), or physical examination findings of typical AF signs including completely irregular cardiac rhythm, variable intensity of the first heart sound, and pulse deficit.
4. Having definite indications for anticoagulant therapy (suspected cardiogenic embolism, e.g., atrial fibrillation, known artificial heart valve, suspected endocarditis, etc.).
5. Patients who have received intravenous thrombolysis, intra-arterial thrombolysis, mechanical thrombectomy, or any revascularization surgery after the current onset, or plan to receive such procedures within 90 days.
6. Use of antiplatelet agents other than aspirin and clopidogrel (e.g., ticagrelor, prasugrel) within 7 days.
7. History of gastrointestinal bleeding, intracranial hemorrhage, massive hemorrhage or blood transfusion in the recent period (excluding mild hemoptysis and mild abnormal vaginal bleeding), or history of other hemorrhagic diseases caused by coagulation dysfunction (e.g., purpura).
8. Having contraindications to or intolerance of clopidogrel, ticagrelor, or aspirin, including:

   * Known history of hypersensitivity;
   * Severe hepatic or renal insufficiency (definition of severe hepatic insufficiency: ALT > 2× upper limit of normal [ULN] or AST > 2× ULN; definition of severe renal insufficiency: creatinine > 1.5× ULN);
   * Severe heart failure (NYHA Class Ⅲ or Ⅳ);
   * Coagulation disorders or history of systemic hemorrhage;
   * History of previous thrombocytopenia or neutropenia;
   * History of previous drug-induced hematological diseases or hepatic dysfunction.
9. Leukopenia (< 2×10⁹/L) or thrombocytopenia (< 100×10⁹/L).
10. Use of heparin or oral anticoagulants within 10 days prior to enrollment.
11. Patients with severe cardiac, pulmonary, hepatic, or renal insufficiency, and those with severe comorbidities (e.g., malignancy, chronic airflow limitation, severe dementia, severe heart failure).
12. Women of childbearing age with a negative pregnancy test but who refuse to adopt effective contraceptive measures; pregnant or lactating women.
13. Poor compliance, unable to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5138 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke (including ischemic and hemorrhagic stroke) within 90 days | within 90 days

SECONDARY OUTCOMES:
Recurrent ischemic stroke | On the 7th day, at 30 days, and within 1 year
New-onset vascular events | On the 7th day, at 30 days, at 90 days and within 1 year.
  Including cardiovascular and cerebrovascular strokes, myocardial infarctions, and vascular deaths.
Modified Rankin Scale (mRS) score | at 30 days, 90 days, and 1 year
  The score range of the scale is from 0 to 6. The higher the score, the worse the outcome.
Recurrent stroke | On the 7th day, the 30th day, the 90th day and within one year.
Worsening of nerve damage (an increase in the NIHSS score by ≥ 4 points compared to the baseline) | At the 24th hour and on the 7th day
Quality of life at day 90 [assessed by the EuroQol - 5 dimension (EQ - 5D) questionnaire] | at 90 days
  It is usually represented by a value between 0 and 1, where 1 represents perfect health, 0 represents death, and the intermediate values reflect different degrees of health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Chen W, Pan Y, Yan H, Meng X, Liu L, Wang Y, Wang Y. Ticagrelor Is Superior to Clopidogrel in Inhibiting Platelet Reactivity in Patients With Minor Stroke or TIA. Front Neurol. 2020 Jun 10;11:534. doi: 10.3389/fneur.2020.00534. eCollection 2020. PMID 32587571
- [Background] Savcic M, Hauert J, Bachmann F, Wyld PJ, Geudelin B, Cariou R. Clopidogrel loading dose regimens: kinetic profile of pharmacodynamic response in healthy subjects. Semin Thromb Hemost. 1999;25 Suppl 2:15-9. PMID 10440417
- [Background] Wang Y, Chen W, Lin Y, Meng X, Chen G, Wang Z, Wu J, Wang D, Li J, Cao Y, Xu Y, Zhang G, Li X, Pan Y, Li H, Zhao X, Liu L, Lin J, Dong K, Jing J, Johnston SC, Wang D, Wang Y; PRINCE Protocol Steering Group. Ticagrelor plus aspirin versus clopidogrel plus aspirin for platelet reactivity in patients with minor stroke or transient ischaemic attack: open label, blinded endpoint, randomised controlled phase II trial. BMJ. 2019 Jun 6;365:l2211. doi: 10.1136/bmj.l2211. PMID 31171523
- [Background] Zhu HC, Li Y, Guan SY, Li J, Wang XZ, Jing QM, Wang ZL, Han YL. Efficacy and safety of individually tailored antiplatelet therapy in patients with acute coronary syndrome after coronary stenting: a single center, randomized, feasibility study. J Geriatr Cardiol. 2015 Jan;12(1):23-9. doi: 10.11909/j.issn.1671-5411.2015.01.003. PMID 25678901
- [Background] Cayla G, Cuisset T, Silvain J, Leclercq F, Manzo-Silberman S, Saint-Etienne C, Delarche N, Bellemain-Appaix A, Range G, El Mahmoud R, Carrie D, Belle L, Souteyrand G, Aubry P, Sabouret P, du Fretay XH, Beygui F, Bonnet JL, Lattuca B, Pouillot C, Varenne O, Boueri Z, Van Belle E, Henry P, Motreff P, Elhadad S, Salem JE, Abtan J, Rousseau H, Collet JP, Vicaut E, Montalescot G; ANTARCTIC investigators. Platelet function monitoring to adjust antiplatelet therapy in elderly patients stented for an acute coronary syndrome (ANTARCTIC): an open-label, blinded-endpoint, randomised controlled superiority trial. Lancet. 2016 Oct 22;388(10055):2015-2022. doi: 10.1016/S0140-6736(16)31323-X. Epub 2016 Aug 28. PMID 27581531
- [Background] Galli M, Benenati S, Capodanno D, Franchi F, Rollini F, D'Amario D, Porto I, Angiolillo DJ. Guided versus standard antiplatelet therapy in patients undergoing percutaneous coronary intervention: a systematic review and meta-analysis. Lancet. 2021 Apr 17;397(10283):1470-1483. doi: 10.1016/S0140-6736(21)00533-X. PMID 33865495
- [Background] Zheng YY, Wu TT, Yang Y, Hou XG, Gao Y, Chen Y, Yang YN, Li XM, Ma X, Ma YT, Xie X. Personalized antiplatelet therapy guided by a novel detection of platelet aggregation function in stable coronary artery disease patients undergoing percutaneous coronary intervention: a randomized controlled clinical trial. Eur Heart J Cardiovasc Pharmacother. 2020 Jul 1;6(4):211-221. doi: 10.1093/ehjcvp/pvz059. PMID 31603191
- [Background] Ma L, Chen W, Pan Y, Yan H, Li H, Meng X, Wang Y, Wang Y. Comparison of VerifyNow, thromboelastography, and PL-12 in patients with minor ischemic stroke or transient ischemic attack. Aging (Albany NY). 2021 Mar 3;13(6):8396-8407. doi: 10.18632/aging.202650. Epub 2021 Mar 3. PMID 33686963
- [Background] Yue C, Lin Z, Lu C, Chen H. Efficacy of Monitoring Platelet Function by an Automated PL-12 Analyzer During the Treatment of Acute Cerebral Infarction With Antiplatelet Medicine. Clin Appl Thromb Hemost. 2021 Jan-Dec;27:10760296211001119. doi: 10.1177/10760296211001119. PMID 33749312
- [Background] Wang Y, Meng X, Wang A, Xie X, Pan Y, Johnston SC, Li H, Bath PM, Dong Q, Xu A, Jing J, Lin J, Niu S, Wang Y, Zhao X, Li Z, Jiang Y, Li W, Liu L, Xu J, Chang L, Wang L, Zhuang X, Zhao J, Feng Y, Man H, Li G, Wang B; CHANCE-2 Investigators. Ticagrelor versus Clopidogrel in CYP2C19 Loss-of-Function Carriers with Stroke or TIA. N Engl J Med. 2021 Dec 30;385(27):2520-2530. doi: 10.1056/NEJMoa2111749. Epub 2021 Oct 28. PMID 34708996
- [Background] Yi X, Lin J, Zhou Q, Wu L, Cheng W, Wang C. Clopidogrel Resistance Increases Rate of Recurrent Stroke and Other Vascular Events in Chinese Population. J Stroke Cerebrovasc Dis. 2016 May;25(5):1222-1228. doi: 10.1016/j.jstrokecerebrovasdis.2016.02.013. Epub 2016 Feb 28. PMID 26935114
- [Background] Wu Y, Shen H, Cai B, Chen C, Yin Q, Zhao Y, Zhou G. Factors associated with clopidogrel resistance and clinical outcomes in ischemic cerebrovascular disease: A retrospective study. J Stroke Cerebrovasc Dis. 2024 Jun;33(6):107684. doi: 10.1016/j.jstrokecerebrovasdis.2024.107684. Epub 2024 Mar 20. PMID 38518890
- [Background] Estevez B, Du X. New Concepts and Mechanisms of Platelet Activation Signaling. Physiology (Bethesda). 2017 Mar;32(2):162-177. doi: 10.1152/physiol.00020.2016. PMID 28228483
- [Background] Franchi F, Rollini F, Angiolillo DJ. Antithrombotic therapy for patients with STEMI undergoing primary PCI. Nat Rev Cardiol. 2017 Jun;14(6):361-379. doi: 10.1038/nrcardio.2017.18. Epub 2017 Feb 23. PMID 28230176
- [Background] Mastenbroek TG, van Geffen JP, Heemskerk JW, Cosemans JM. Acute and persistent platelet and coagulant activities in atherothrombosis. J Thromb Haemost. 2015 Jun;13 Suppl 1:S272-80. doi: 10.1111/jth.12972. PMID 26149036
- [Background] Gao Y, Chen W, Pan Y, Jing J, Wang C, Johnston SC, Amarenco P, Bath PM, Jiang L, Yang Y, Wang T, Han S, Meng X, Lin J, Zhao X, Liu L, Zhao J, Li Y, Zang Y, Zhang S, Yang H, Yang J, Wang Y, Li D, Wang Y, Liu D, Kang G, Wang Y, Wang Y; INSPIRES Investigators. Dual Antiplatelet Treatment up to 72 Hours after Ischemic Stroke. N Engl J Med. 2023 Dec 28;389(26):2413-2424. doi: 10.1056/NEJMoa2309137. PMID 38157499
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Liu L, Wang D, Wong KS, Wang Y. Stroke and stroke care in China: huge burden, significant workload, and a national priority. Stroke. 2011 Dec;42(12):3651-4. doi: 10.1161/STROKEAHA.111.635755. Epub 2011 Nov 3. PMID 22052510
- [Background] Wang W, Jiang B, Sun H, Ru X, Sun D, Wang L, Wang L, Jiang Y, Li Y, Wang Y, Chen Z, Wu S, Zhang Y, Wang D, Wang Y, Feigin VL; NESS-China Investigators. Prevalence, Incidence, and Mortality of Stroke in China: Results from a Nationwide Population-Based Survey of 480 687 Adults. Circulation. 2017 Feb 21;135(8):759-771. doi: 10.1161/CIRCULATIONAHA.116.025250. Epub 2017 Jan 4. PMID 28052979
- [Background] Tu WJ, Zhao Z, Yin P, Cao L, Zeng J, Chen H, Fan D, Fang Q, Gao P, Gu Y, Tan G, Han J, He L, Hu B, Hua Y, Kang D, Li H, Liu J, Liu Y, Lou M, Luo B, Pan S, Peng B, Ren L, Wang L, Wu J, Xu Y, Xu Y, Yang Y, Zhang M, Zhang S, Zhu L, Zhu Y, Li Z, Chu L, An X, Wang L, Yin M, Li M, Yin L, Yan W, Li C, Tang J, Zhou M, Wang L. Estimated Burden of Stroke in China in 2020. JAMA Netw Open. 2023 Mar 1;6(3):e231455. doi: 10.1001/jamanetworkopen.2023.1455. PMID 36862407
- [Background] Tu WJ, Wang LD; Special Writing Group of China Stroke Surveillance Report. China stroke surveillance report 2021. Mil Med Res. 2023 Jul 19;10(1):33. doi: 10.1186/s40779-023-00463-x. PMID 37468952